CLINICAL TRIAL: NCT01564069
Title: Intrathecal Therapy for Chronic Non-Cancer Pain: An Analysis of Its Efficacy
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Srdjan Nedeljkovic, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2007P000874
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Intrathecal pain management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- IT opioids: Patients with IT pumps receiving IT opioids
- Systemic opioids: Patients taking oral or transdermal opioids for chronic pain
- Non-opioid management: Patients managing chronic pain without taking opioids

SUMMARY:
Our hypothesis is that patients with intrathecal delivery systems for chronic non-cancer pain will report no improvement treatment efficacy when compared to patients with chronic pain managed with oral or systemic opioid therapies. Our secondary hypothesis is that patients with intrathecal delivery systems for chronic non-cancer pain will report no improvement in treatment efficacy when compared to patients with chronic pain who are managed with non-opioid therapies.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 18 years of age with legal decision making ability.
* Subjects receiving care at the Brigham and Women's Hospital Pain Management Center.
* Subjects must have a history of chronic pain > 6 months and must have been a patient in the BWH Pain Center > 6 months.

Exclusion Criteria:

* Pain due to metastatic cancer or to cancer that is locally invasive
* Patients with a primary diagnosis of spasticity, receiving intrathecal baclofen
* Evidence of psychosis or hospitalization for psychiatric illness during study
* Pregnancy at any time during the study
* Altered mental status that would make subject unable to complete outcome questionnaires
* Significant chronic medical illness, such that requires frequent hospitalization or health care utilization (ie: renal failure requiring dialysis, heart failure or cardiac disease requiring surgery or intensive care admission, pulmonary disease requiring intubation or hospitalization, pancreatitis requiring hospitalization, vascular disease requiring surgery or hospitalization, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females greater than 18 years of age History of chronic pain greater than 6 months Patient in the BWH Pain Center for greater than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-03-31 (Actual)

PRIMARY OUTCOMES:
Treatment Efficacy of Intrathecal Infusions | March 2014
  The primary objective of this study is to evaluate the treatment efficacy of intrathecal infusions for chronic pain and compare this form of therapy to systemic opioid therapy and non-opioid therapy for chronic pain > 6 months duration.

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan S Nedeljkovic, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States